CLINICAL TRIAL: NCT01856946
Title: Effect of 4,000 IU Vitamin D3 Supplementation on Oral Glucose Tolerance Among Vitamin D Deficient Obese Adolescent
Brief Title: Effect of Vitamin D Supplementation on Oral Glucose Tolerance Among Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Aneesh Tosh, Associate Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1203853
Record Dates: First submitted 2013-05-10; First posted 2013-05-20 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4,000 IU Vitamin D3 (Experimental): two 2,000 IU vitamin D3 pills (total 4,000 IU) daily for six months.
  Interventions: Dietary Supplement: 4,000 IU vitamin D3

INTERVENTIONS:
Dietary Supplement: 4,000 IU vitamin D3 — two 2,000 IU vitamin D3 pills (total 4,000 IU) daily for six months.

SUMMARY:
Childhood obesity is a rapidly growing epidemic in the US and the world. Current estimates suggest that 30% of our nation's children are either overweight ot obese. Obesity is a major risk factor towards the development of insulin resistance, which, in turn is a major risk factor for the development of type 2 diabetes. Prior research has suggested that vitamin D therapy may be a safe, inexpensive, and effective method of reducing insulin resistance and a person's risk of developing diabetes.

The investigators' prior studies have shown that daily 4,000 IU vitamin D therapy is a safe and effective method of improving insulin resistance based on a calculation called the HOMA-IR.

The next step in identifying whether vitamin D truly improves insulin resistance is to use oral glucose tolerance testing (OGTT), which is a better real-life measure of insulin resistance compared to the previously used HOMA-IR.

DETAILED DESCRIPTION:
The investigators intend to recruit 20 obese adolescent subjects from the PI's obesity clinic to participate in the study. Investigators expect 5 to drop out, therefore leaving 15 subjects to complete the study. Eligible and assenting subjects (with consent from a parent) will be admitting to the Pediatric Procedure Suite and MU Women's and Children's Hospital. They will have an IV placed in the arm by a nurse experienced with working with children. The subjects will have blood drawn from the IV checking for vitamin D level, insulin, glucose, and c-peptide level (another marker for insulin status). The subject will then be asked to drink a 75 gram glucose solution. Additional blood will be drawn from the IV site to check for glucose, insulin, and c-peptide levels at 30 minutes, 60 minutes, 90 minutes, and 120 minutes. A total of 30 mL (2 tablespoons) of blood will be drawn that day. The subject will have the IV removed and will be discharged to then take two 2,000 IU vitamin D3 pills (total 4,000 IU) daily for six months.

At a routine 3 months clinical visit, the subject will be tested for routine, standard of care, basic metabolic profile (BMP) with 4 ml of blood (less than 1 teaspoon) to assess for high calcium levels, a potential complication of vitamin D therapy. In the investigators' previous study of adolescents taking 4,000 IU vitamin D daily for six months, no subject developed a high calcium level.

At six months, the subject will return to the Pediatric procedure suite to have another OGTT and labs via IV as described above.

ELIGIBILITY:
Inclusion Criteria:

* Obese adolescent (BMI >85th percentile for age)
* 9-19 years of age
* attending the ADOBE clinic at the University of Missouri
* 25OH vitamin D level within past 3 months

Exclusion Criteria:

* use of vit D supplements other than standard multi-vitamin preparation (i.e., should not be receiving vit D > 1000 IU/d)
* use of medications that interfere with vit D metabolism (e.g., anti-convulsive)
* history of hepatic or renal disorders, hypercalciuria, or hypercalcemia
* undergoing UV radiation as medical therapy
* pregnancy; cigarette smoking; current use of a tanning bed
* current type 2 diabetes
* any current antihyperglycemic medication use (e.g. metformin, insulin) less than one month prior to initial OGTT.

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
change in oral glucose tolerance | baseline and 6 months
  Will obtain oral glucose tolerance tests at baseline and at 6 months to determine change

CONTACTS AND LOCATIONS:
Overall Officials: Aneesh K Tosh, MD. MS, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Adolescent Obesity Clinic, Columbia, Missouri, United States

REFERENCES:
- [Background] Belenchia AM, Tosh AK, Hillman LS, Peterson CA. Correcting vitamin D insufficiency improves insulin sensitivity in obese adolescents: a randomized controlled trial. Am J Clin Nutr. 2013 Apr;97(4):774-81. doi: 10.3945/ajcn.112.050013. Epub 2013 Feb 13. PMID 23407306